CLINICAL TRIAL: NCT06061705
Title: Identification of Individual Histological and Blood Markers in Patients With Recurrent or Metastatic Upper Aerodigestive Tract Squamous Cell Carcinoma in Response to Immunotherapies
Acronym: iMonitORL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: iMonitORL
Record Dates: First submitted 2023-09-11; First posted 2023-09-29 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- procedure/surgery: Tumor biopsy (Experimental): Following the start of immunotherapy, an ENT surgeon will perform a cervico-facial tumor biopsy between D30 and D180.
  Interventions: Procedure: Tumor Biopsy

INTERVENTIONS:
Procedure: Tumor Biopsy — Following the start of immunotherapy, an ENT surgeon will perform a cervico-facial tumor biopsy between D30 and D180. This will only be carried out if the tumour tissue is externalized and therefore accessible, and if the biopsy can be performed under local anaesthetic without any constraints for the patient (pain, risk of bleeding).
  It consists of a superficial sampling of the externalized tumour lesion under local anaesthetic (xylocaine spray 5%, or xylocaine injectable 1%).
  Biopsy of cervico-facial lesions under local anaesthetic is a commonly performed procedure. The main risk of this procedure is bleeding, which is very rare.
  The biopsy will not be performed if the surgeon considers that the risk of bleeding is too great. Given the externalized nature of the lesion, biopsy does not entail any risk of tumour dissemination (possible for deep biopsies).
  * Four 10-mL blood samples from two heparinized tubes
  * Four 5-mL unstimulated saliva samples: non-invasive examination.

SUMMARY:
Epidermoid Carcinoma of the Upper Aerodigestive Tract (CEVADS) is the 6th most common cancer worldwide. Despite current therapies (radiotherapy, surgery and chemotherapy), cancers of the Upper Aerodigestive Tract (UAT) have a poor prognosis, with a 10-year survival rate of no more than 20%.

For recurrent or metastatic CEVADS, the therapeutic arsenal, based for many years on chemotherapy and anti-EGFR (Epidermal Growth Factor Receptor) agents, has been enriched by a new therapeutic class: PD-1 inhibitors. For CEVADS, PD-1 inhibitors have been approved for second-line treatment of nivolumab for over a year, and are now used in first-line treatment of pembrolizumab.

The results of this therapeutic class in CEVADS are not as spectacular as for melanoma or bronchial cancer. Indeed, only 20% of patients have a favorable response, compared with half who experience disease progression. This low proportion of responders can be explained by tumor heterogeneity within CEVADS and poor patient selection.

The only marker used to select patients is PD-L1 expression detected by ImmunoHistochemistry (IHC). However, it seems that this marker, described as imperfect, is still little explored in ENT. It needs to be compared with the expression of other cell lines in the tumor microenvironment, which could play an important role in resistance to PD-1 inhibitors.

IHC identifies all macrophages using the CD68 marker, while the CD163 marker is specific to M2 macrophages.

Other targets in the microenvironment are also being investigated, with the discovery of a Tertiary Lymphocyte Structure (TLS) in melanoma treated with immunotherapy.

It therefore seems necessary to gain a better understanding of the mechanisms of tumor progression under immunotherapy in order to develop strategies to optimize response to treatment. This would enable better selection of patients likely to benefit from immunotherapy, and open up prospects for therapeutic combinations.

The hypothesis is that macrophages, but also other cells and factors in the CEVADS microenvironment, play a decisive role in resistance to PD-1 inhibitors. The aim is therefore to continue these macrophage analyses, extend them to other cells in the microenvironment and link them to other prognostic factors under investigation.

A prospective study will analyze tumor tissue during treatment with PD-1 inhibitors, in order to correlate all the factors studied with response or resistance to immunotherapies.

In addition, the oral microbiota, in the lineage of the intestinal microbiota, has been shown to be highly stable over time and to play a role in the oncogenesis of certain cancers, notably CEVADS. Like the intestinal microbiota, it could also represent a prognostic factor in the response to immunotherapies.

Of all the bacteria in this oral microbiota, one has been shown to play a major role: Fusobacterium nucleatum (F. nucleatum). However, little is known about the mechanism of action of intratumoral F. nucleatum on the development of CEVADS. In particular, it is thought to play a role in local cancer immunity, via macrophages, regulatory T cells (Tregs) and TLRs. Finally, it appears that specific antimicrobial T-cell responses may cross-react with tumor antigens, hence the importance of also analyzing the metabolome of commensal bacteria.The aim of this study was to evaluate the evolution of the presence of this bacterium in saliva, as well as the specific immune response to F. nucleatum in patients with CEVADS during immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with histologically confirmed CEVADS involving the oral cavity, oropharynx, hypopharynx or larynx
* Pre-treated patients with a first recurrence (locoregional or metastatic) who are candidates for immunotherapy
* Patient affiliated to a health insurance plan
* French-speaking patient
* Patient with free, informed and written consent

Exclusion Criteria:

* Patients with a contraindication to immunotherapy (transplant patients)
* Pregnant or breast-feeding patients
* Patient under guardianship or curatorship
* Patient under court protection
* Patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Histological markers linked to the clinical benefit of immunotherapies | Month 6
  This outcome corresponds to the number of patients presenting a clinical benefit: objective response or stable disease according to RECIST v1.1 dimensional criteria, and the number of patients presenting tumor progression as the best response to immunotherapy.

SECONDARY OUTCOMES:
Histological markers linked to survival | Month 6
  This outcome corresponds to the time elapsed between initiation of immunotherapy and death, all causes combined.
Expression of histological markers with PD-L1 expression | Month 6
  This outcome corresponds to the quantitative or semi-quantitative evolution of each marker including incidence of macrophages, lymphocytes, epithelial-mesenchymal transition markers) and blood (including Squamous Cell Carcinoma (SCC), neutrophil/lymphocyte ratio, circulating macrophages and lymphocytes), compared with the quantitative evolution of PD-L1 expression.
Presence of Fusobacterium nucleatum in the oral microbiota | Month 6
  This outcome corresponds to the presence of Fusobacterium nucleatum in the oral microbiota by microbial DNA detection.
Presence of an IgG or IgA anti-Fusobacterium nucleatum humoral response | Month 6
  This outcome corresponds to the presence of an anti-F. nuc IgG or IgA humoral response in patients' serum before and after immunotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Raymond, MD, PhD, Study Director — Hôpital Paris Saint-Joseph
Locations (3):
- France (3):
  - Hôpital Saint-Joseph, Paris
  - Hôpital Bichat, Paris
  - Hôpital Saint-Louis, Paris

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Cohen EEW, Soulieres D, Le Tourneau C, Dinis J, Licitra L, Ahn MJ, Soria A, Machiels JP, Mach N, Mehra R, Burtness B, Zhang P, Cheng J, Swaby RF, Harrington KJ; KEYNOTE-040 investigators. Pembrolizumab versus methotrexate, docetaxel, or cetuximab for recurrent or metastatic head-and-neck squamous cell carcinoma (KEYNOTE-040): a randomised, open-label, phase 3 study. Lancet. 2019 Jan 12;393(10167):156-167. doi: 10.1016/S0140-6736(18)31999-8. Epub 2018 Nov 30. PMID 30509740
- [Background] Leemans CR, Snijders PJF, Brakenhoff RH. The molecular landscape of head and neck cancer. Nat Rev Cancer. 2018 May;18(5):269-282. doi: 10.1038/nrc.2018.11. Epub 2018 Mar 2. PMID 29497144
- [Background] Evrard D, Hourseau M, Couvelard A, Paradis V, Gauthier H, Raymond E, Halimi C, Barry B, Faivre S. PD-L1 expression in the microenvironment and the response to checkpoint inhibitors in head and neck squamous cell carcinoma. Oncoimmunology. 2020 Nov 19;9(1):1844403. doi: 10.1080/2162402X.2020.1844403. PMID 33299655
- [Background] Wondergem NE, Nauta IH, Muijlwijk T, Leemans CR, van de Ven R. The Immune Microenvironment in Head and Neck Squamous Cell Carcinoma: on Subsets and Subsites. Curr Oncol Rep. 2020 Jun 29;22(8):81. doi: 10.1007/s11912-020-00938-3. PMID 32602047
- See also: SEER Cancer Statistics Review (CSR) 1975-2014 — https://seer.cancer.gov/archive/csr/1975_2014/